CLINICAL TRIAL: NCT01295047
Title: Effects of Atenolol, Perindopril and Verapamil on Haemodynamic and Vascular Function in Marfan Syndrome - A Randomised Double-Blind Crossover Trial
Brief Title: Comparison of Medical Therapies in Marfan Syndrome.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: DR ALAN FRASER, WALES HEART RESEARCH INSTITUTE
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPONCU101; 2005-000749-13 (EudraCT Number)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2006-01

CONDITIONS: Marfan Syndrome
Keywords: Marfan Syndrome; Large arterial function; LV function; atenolol; perindopril; verapamil; central arterial pressure
MeSH Terms: conditions — Marfan Syndrome | interventions — Atenolol; Verapamil; Perindopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ATENOLOL (Active Comparator): ATENOLOL 75MG FOR 4 WEEKS
  Interventions: Drug: Atenolol
- VERAPAMIL (Active Comparator): 240MG VERAPAML FOR 4 WEEKS
  Interventions: Drug: VERAPAMIL
- PERINDOPRIL (Active Comparator): 4MG PERINDOPRIL FOR 4 WEEKS
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: Atenolol
  Arms: ATENOLOL
Drug: VERAPAMIL — 240 MG SR
  Arms: VERAPAMIL
Drug: Perindopril — 4 MG
  Arms: PERINDOPRIL

SUMMARY:
The investigators are looking at the different impacts of atenolol, verapamil and perindopril on large artery and lv function in marfan syndrome. It is a double-blind, randomised cross-over trial.

DETAILED DESCRIPTION:
The investigators recruited 21 patients with confirmed diagnosis of Marfan syndrome from two centres. The investigators performed radial artery applanation tonometry and pulse wave analysis to derive central aortic pressure and haemodynamic indexes pre-and post administering Atenolol 75mg, Perindopril 4mg and Verapamil 240mgs each for four weeks with a two week wash-out between medications. All patients underwent detailed functional and anatomical echocardiographic assessments at each visit.

Inclusion criteria were ages 16-60 years with no treatment or β-blocker or other monotherapy only for Marfan syndrome. Patients with previous aortic dissection or aortic surgery, severe valvular regurgitation, aortic diameter at the sinotubular junction ≥ 5.0cm, contraindications to specific drug treatment, e.g. asthma and β-blocker, or those who were pregnant or at risk of pregnancy were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16-60 years old with no treatment or β-blocker or other monotherapy only for Marfan syndrome

Exclusion Criteria:

* Previous aortic dissection or aortic surgery
* Severe valvular regurgitation
* Aortic diameter at the sinotubular junction ≥ 5.0cm
* Contraindications to specific drug treatment, e.g. asthma and β-blocker
* Those who were pregnant or at risk of pregnancy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
CENTRAL ARTERIAL PRESSURE | 18 weeks
  CENTRAL ARTERIAL PRESSURE MEASURED BY APPLANATION TONOMETRY

SECONDARY OUTCOMES:
LARGE ARTERIAL STIFFNESS INDICES | 18 WEEKS
  MEASURED BY ECHO AND BY PULSE WAVE VELOCITY/ANALYSIS BY APPLANATION TONOMETRY
LV Function | 18 WEEKS
  GLOBAL AND REGIONAL MARKERS BY ECHO

CONTACTS AND LOCATIONS:
Locations (1):
- Wales Heart Research Institute, Cardiff University, Cardiff, United Kingdom